CLINICAL TRIAL: NCT00394303
Title: Tight Intra-Operative Glucose Control Using Continuous Insulin Infusion During Coronary Artery Bypass Surgery: Randomized Controlled Trial
Brief Title: Tight Intra-Operative Glucose Control During Coronary Artery Bypass Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Trial suspended on 26 February, following the publication of a trial with negative results (Ann Intern Med 146(4), 2007). Pending ethics committee re-approval.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Dr. Mical Paul, Rabin Medical Center, Beilinson Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4214
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2007-06

CONDITIONS: Coronary Artery Bypass
Keywords: Open heart surgery; Diabetes mellitus; Hyperglycemia; Surgical site infection; Normoglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention
  Interventions: Drug: Intraoperative continuous insulin infusion
- 2 (No Intervention): Control
  Interventions: Other: Control

INTERVENTIONS:
Drug: Intraoperative continuous insulin infusion — Nomogram specified in appendix
  Arms: 1
Other: Control — Glucose management according to the discretion of the anesthesiologist aimed to maintain glucose levels <200 mg.dl, reflecting current practice.
  Arms: 2

SUMMARY:
Blood glucose levels increase in response to stress, infection or other conditions faced by patients in the hospital. This occurs commonly among patients with known diabetes, but also among non-diabetic hospitalized patients. Tight glucose control, the maintenance of blood glucose levels within normal limits (80-120 mg/dl), has been shown to improve patient outcomes in the hospital in several settings, mainly among critically ill patients hospitalized in intensive care units.

We plan to assess the importance of tight glucose control during open-heart surgery. The prevalence of hyperglycemia (elevated blood glucose) during this operation is high. Hyperglycemia may be associated with increased vulnerability to surgical site infections, neurological damage, cardiac and renal injury. Conversely, tight glucose control may be associated with hypoglycemia (pathologically low glucose levels) that may results in neurological injury. We hypothesize that tight glucose control will improve patient outcomes following surgery.

DETAILED DESCRIPTION:
Current evidence supports intensive glucose control for patients in the intensive care unit post-cardiac surgery. The risk-benefit ratio of tight glucose control using continuous insulin infusion during surgery has not been established. Pros for tight control include the association of hyperglycemia with neurological injury, cardiac ischemia, white blood cell dysfunction and renal failure. The cons include adverse effects, mainly hypoglycemia and hypokalemia. As with any intervention in medicine, tight intra-operative glucose control should be assessed in a randomized controlled trial.

Objectives:to assess whether tight intra-operative tight glucose control using continuous insulin infusion reduces morbidity and mortality following cardiac surgery, defined as the incidence rate of surgical site infections, adverse neurological events, renal failure and 30-day mortality following CABG.

Additional outcomes will include the effect of continuous insulin infusion on longer-term mortality; other infectious complications and antibiotic use during hospitalization; cardiovascular outcomes; the need for re-operations; length of hospital stay; readmission; hypoglycemia and other adverse events.

Design: randomized controlled trial, with blinding of outcome assessors.

Participants: all consecutive patients >18 years undergoing CABG, without or without additional valve or other surgery at Rabin Medical Center; Beilinson campus, providing informed consent.

Exclusion criteria: patients with diabetic ketoacidosis, or hyperosmolar coma.

Intervention: Continuous insulin infusion throughout the operation aimed to maintain normoglycemia using a nomogram

Control: Glucose management according to the discretion of the anesthesiologist (continuous or bolus infusion)

During the early post-operative period (ICU-stay following surgery), all patients will be treated with intensive glucose control targeting glucose levels between 80-110.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients >18 years undergoing CABG, without or without additional valve or other surgery at Rabin Medical Center; Beilinson campus, providing informed consent.

Exclusion Criteria:

* Patients with diabetic ketoacidosis, or hyperosmolar coma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2007-02; Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality. | 30-day
Deep or organ/ space (mediastinitis) surgical site infections. | 90 days
Acute renal failure during post-operative ICU stay, defined as: doubling of serum creatinine from baseline; or >50% reduction from baseline glomerular filtration rate; or need for renal replacement therapy. | 30 days
Perioperative cerebrovascular event defined as any new, temporary or permanent, focal or global neurological deficit. | 30 days

SECONDARY OUTCOMES:
Individual components of the composite primary outcome | 30 days
6-months and long-term survival. | 6 ans 12 months
Other infectious complications during ICU stay including pneumonia and bloodstream infections according to CDC criteria | ICU stay
Antibiotic use | 30 days
Durations of intubation, ICU and hospital stay | hospital stay
Other post-operative complications occurring during ICU stay, including re-intubation, re-operation | ICU stay
Occurrence of hypoglycemia, defined as blood glucose level of 50mg/ dl or less, during surgery and up to the first glucose measurement in ICU. | during surgery
Occurrence of severe hypokalemia, defined as K<2.5 mEq/l, during surgery | during surgery
Glucose control in ICU, during the first 2 post-operative days | 2 post-operative days
Neurological status before surgery, at discharge and 3 months following surgery: | 3 months
Adverse cardiac events occurring during ICU stay | ICU stay
Re-hospitalizations | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mical Paul, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikvah, Israel